CLINICAL TRIAL: NCT05482113
Title: Opioid Consumption in Patients Undergoing Arthroscopic Rotator Cuff Repair Using Interscalene Brachial Plexus Blocks With and Without Liposomal Bupivacaine: A Randomized Controlled Trial
Brief Title: Measuring Opioid Use After Rotator Cuff Repair: Comparing the Effects of Standard vs. Extended-release Nerve Blocks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Carilion Clinic (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Thomas K Miller, M.D., Section Chief, Sports Medicine, Carilion Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-530
Record Dates: First submitted 2021-07-20; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Rotator Cuff Tears
Keywords: randomized controlled trial; exparel; opioid use; arthroscopic rotator cuff repair; bupivacaine; liposomal bupivacaine; rotator cuff; interscalene brachial plexus block; rotator cuff tear
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control - Standard Bupivacaine (Active Comparator): After proper positioning and local infiltration, a linear high-frequency ultrasound transducer will be placed on the anteromedial aspect of the neck, approximately 2 cm above the clavicle, and the interscalene brachial plexus will be identified between the anterior and middle scalene muscles. After sterile preparation of the skin, a 22-gauge needle will be inserted in-plane from the lateral aspect of the transducer and directed through the middle scalene muscle. The needle will be advanced until the tip is observed just lateral to the brachial plexus sheath. After negative aspiration, 20mL of 0.5% bupivacaine will be injected in 5mL increments, followed by 20mL of 0.25% bupivacaine injected in 5mL increments. The injection will be administered slowly with periodic aspiration, with the needle being adjusted using ultrasound guidance as the ISB is injected to surround the brachial plexus trunks (upper, middle and lower) that are seen at the interscalene level of injection.
  Interventions: Drug: Bupivacaine Hcl 0.25% Inj
- Experimental - Liposomal Bupivacaine (Exparel) (Experimental): After proper positioning and local infiltration, a linear high-frequency ultrasound transducer will be placed on the anteromedial aspect of the neck, approximately 2 cm above the clavicle, and the interscalene brachial plexus will be identified between the anterior and middle scalene muscles. After sterile preparation of the skin, a 22-gauge needle will be inserted in-plane from the lateral aspect of the transducer and directed through the middle scalene muscle. The needle will be advanced until the tip is observed just lateral to the brachial plexus sheath. After negative aspiration, 20mL of 0.5% bupivacaine will be injected in 5mL increments, followed by 20mL of Exparel injected in 5mL increments. The injection will be administered slowly with periodic aspiration, with the needle being adjusted using ultrasound guidance as the ISB is injected to surround the brachial plexus trunks (upper, middle and lower) that are seen at the interscalene level of injection.
  Interventions: Drug: Liposomal bupivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine — Liposomal Bupivacaine (Exparel) Brachial Plexus Block for Arthroscopic Rotator Cuff Repair
  Other Names: Exparel
  Arms: Experimental - Liposomal Bupivacaine (Exparel)
Drug: Bupivacaine Hcl 0.25% Inj — Standard 0.25% Bupivacaine Brachial Plexus Block for Arthroscopic Rotator Cuff Repair
  Other Names: Standard Bupivacaine
  Arms: Control - Standard Bupivacaine

SUMMARY:
The investigators aim to determine if a longer acting nerve block, which is a local anesthetic, can help reduce opioid use after surgery in patients that are getting rotator cuff repair surgery. The investigators will also determine if the longer acting block can reduce the number of days that opioids are taken after surgery. Patients that schedule this type of surgery will be given information regarding the study and asked if they want to participate. If they do, they will be randomized to either receive the standard nerve block or the longer acting nerve block. Participants and physicians will not know which nerve block the participants are receiving. Participants will receive a standard pain medication prescription after surgery and will be asked to record pain scores, medications taken and satisfaction level every day in a journal for two weeks. Participants will be asked to bring in their medication bottles and pain journal to the 2-week follow up appointment. Participants' pain scores will be assessed in the office at the follow up appointment and study staff will conduct a pill count. Participants will return for a 6-week follow up appointment and pain scores will be assessed again at that time, and another pill count will be conducted. At this point the study will be complete.

DETAILED DESCRIPTION:
1. Patients who have an Arthroscopic Rotator Cuff Repair (ARCR) scheduled to be performed at Roanoke Ambulatory Surgery Center (RASC) by one of the participating surgeons will be prescreened, assessed for eligibility and consented at the pre-operative visit.

   * This office visit already includes: a formatted discussion regarding the risks, benefits and alternatives to surgery; fitting for a sling; and a review of the opioid policy and patient agreement used by Carilion Clinic's Institute for Orthopaedics and Neurosciences (ION).
   * The PI or sub-investigators will conduct the discussion regarding the rational and use of Interscalene Brachial Plexus Block (ISB) with the procedure, the rationale for assessment of alternate medications used for the study and any other pertinent details. An approved research team member will review all sections of the IRB approved research consent in detail, in person at the pre-operative visit. All questions will be answered and physical signatures will be obtained. Both research groups, control and experimental, will sign the same consent document. A copy of the signed consent will be provided to the participant.
2. All participants will be given a pain diary to take home and begin filling out the day following their surgery. Per participant preference, pain diary may be physical copy or done electronically via REDCap.

   - All participants will be instructed on how to record entries in the pain diary by an approved research team member. The pain diary will have templated pages with areas to record the amounts and names of medications they consumed, their Numerical Rating Scale (NRS) score, their Intervention Based Pain Scale (IBPS) score, as well as satisfaction levels and a place to record how long their anesthetic block lasted.
3. Participants in both study groups will be provided the same information and education regarding postoperative pain management protocol and expectations. This includes:

   * A review of the opioid policy and patient agreement used by Carilion Clinic's ION as well as a discussion about proper use of the pain medication to be prescribed for postoperative pain management
   * A discussion regarding the ISBs used with the procedure and their likely duration of analgesia
   * A discussion of scheduled postoperative visits and how to contact the office with questions/concerns regarding recovery
4. The investigators will use the random number generator feature in REDcap to randomly assign subjects to receive the standard Bupivacaine HCl ISB or the Exparel ISB. Surgery schedules at RASC are released on Friday the week before. The investigators will retrieve the surgery schedule on Fridays from RASC, find study subjects, and randomize them to group A (Exparel) or group B (Bupivacaine HCl) that same day (the Friday before surgery). Once the subjects are randomized, the investigators will communicate the randomization to a RASC staff member and they will put the arm designation (group A or group B) in an envelope and attach it to the subject's chart for the day of surgery. The contents of the envelope will only be seen by Anesthesia providers and charge nurses prior to the surgery with no other study staff in the room (so the blind is not broken). Charge nurses and anesthesiologists at RASC will be unblinded to the definitions of groups A & B to gather and administer the proper medications. Surgeons will not be in the room at the time of anesthetic administration. The patient and all other providers including physicians and physician assistants will be blinded to the result of the randomization. Participants may opt to be unblinded to their group assignment at their 6-week post operative visit.
5. All participants will be undergoing a routine ARCR. The procedure will not deviate from the standard of care operation that is typically performed. All participants will receive an ultrasound-guided ISB by a pool of anesthesia providers at RASC. The only difference between subject groups is that the control group will receive a standard Bupivacaine HCl ISB and the experimental group will receive an Exparel ISB.
6. On the day of surgery all participants will be brought to the pre-operative holding area at RASC where they are seen prior to the surgical procedure by both the operating surgeon and the anesthesiologist. The operating surgeon will review the surgical procedure with all participants and will mark the side and location of the procedure. The anesthesiologist will review the ISB procedure with the participant and ensure correct side and location marked by physician. Before the anesthesiologist begins administration of the ISB, an anesthesia time-out is performed with the anesthesiologist and the participant to confirm patient identity, surgical site, and planned procedure.
7. In the pre-operative holding area or the operating room, the anesthesiologist will position all participants in the recumbent position with a slight roll onto the opposite side from the block and will administer a local infiltration of the skin with 1-2mL of Bupivacaine HCl 0.5% (dosages may vary based on participant size and pain threshold). If participants are unable to sit still during ISB administration, they may be sedated by the anesthesiologist with one of the following (Medications and dosages vary based on need):

   * Versed
   * Fentanyl
   * Propofol
8. Administration of the standard Bupivacaine HCl ISB for the control arm goes as follows:

   - After proper positioning and local infiltration, a linear high-frequency ultrasound transducer will be placed on the anteromedial aspect of the neck, approximately 2 cm above the clavicle, and the interscalene brachial plexus will be identified between the anterior and middle scalene muscles. After sterile preparation of the skin, a 22-gauge block needle will be inserted in-plane from the lateral aspect of the transducer and directed through the middle scalene muscle. The needle will be advanced until the tip is observed just lateral to the brachial plexus sheath. After negative aspiration, 20mL of 0.5% bupivacaine will be injected in 5mL increments, followed by 20mL of 0.25% bupivacaine injected in 5mL increments. The injection will be administered slowly with periodic aspiration, with the needle being adjusted using ultrasound guidance as the ISB is injected to surround the brachial plexus trunks (upper, middle and lower) that are seen at the interscalene level of injection. There will be only one injection site.
9. Administration of the Exparel ISB for the experimental arm goes as follows:

   - After proper positioning and local infiltration, a linear high-frequency ultrasound transducer will be placed on the anteromedial aspect of the neck, approximately 2 cm above the clavicle, and the interscalene brachial plexus will be identified between the anterior and middle scalene muscles. After sterile preparation of the skin, a 22-gauge block needle will be inserted in-plane from the lateral aspect of the transducer and directed through the middle scalene muscle. The needle will be advanced until the tip is observed just lateral to the brachial plexus sheath. After negative aspiration, 20mL of 0.5% bupivacaine will be injected in 5mL increments, followed by 20mL of Exparel injected in 5mL increments. The injection will be administered slowly with periodic aspiration, with the needle being adjusted using ultrasound guidance as the ISB is injected to surround the brachial plexus trunks (upper, middle and lower) that are seen at the interscalene level of injection. There will be only one injection site.
10. 15-20 minutes after administration of ISBs (Bupivacaine HCl or Exparel), all participants will be put under general anesthesia (if not already) by the anesthesiologist with one of the following (Medications and dosages vary based on patient need. Most common medications used listed below):

    * Versed
    * Fentanyl
    * Propofol
11. After general anesthetic takes effect, all participants will be operated on by their fellowship-trained orthopaedic surgeon.

    - During the operation, all participants may receive an intravenous injection of Toradol (15-30 mg based on weight and renal function)
12. All participants will be discharged with post-operative pain medications regimens based on department protocol and physician preference.

    * Oral Opioid Medication: 5mg/325mg hydrocodone/acetaminophen q4-6h prn pain
    * Non-Opioid Pain Medication: 10mg Toradol q8h prn pain 5 days maximum
13. All participants will be called or seen in the office within 72 hours after surgery to assess pain status, ensure adequate pain management and will be reminded to complete the pain diary.
14. All participants will fill out a pain diary during the first 2 weeks postoperatively that will assess 5 measures.

    * Medication consumption (dose & number of pills) - will be asked to record daily
    * Pain score on the NRS - will be asked to record daily
    * Pain score on an institutional IBPS - will be asked to record daily
    * Patient satisfaction - will be asked to record daily
    * Nerve block duration - will be reminded to record if their block has worn off, and if so, how many hours it was effective (until they regained sensation).
15. All participants will be called before their 2- and 6-week follow-up appointments and will be asked to bring in their pain diaries as well as their opioid medication pill bottles to their visit so that pill counts may be conducted.

    - All calls will be made by trained, authorized site delegates. There will be a locked drop-box in the ION building where participants can drop off their pain diaries after their 2-week follow-up appointment if they forget to bring it in to their appointment.
16. All participants will come into the office for 2 follow up appointments, at 2 and 6 weeks postoperatively.

    * At the 2-week postoperative visit, all participants will be expected to bring in their opioid medication pill bottles and pain diaries per instructions given at study enrollment and on the reminder phone call. All participants will be shown where the lock boxes are to deposit pain diaries. Pill counts will be conducted and recorded as well as number of refills.
    * At the 6-week postoperative visit, all participants will be expected to bring in the opioid medication pill bottles per instructions given at study enrollment and on the reminder phone call.
    * Pill counts will be conducted and recorded as well as number of refills.
17. All participant follow-up appointments will be conducted at Carilion's Institute for Orthopaedics and Neurosciences (ION) or via telemedicine, and should not take significantly longer than normal follow up appointments. Slightly increased visit duration related to conducting pill counts should not exceed about 5 minutes. All participants will be enrolled in the study for 6 weeks after their surgical date, at which point their involvement in the study will conclude.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age at time of enrollment
2. Be scheduled for Arthroscopic Rotator Cuff Repair (ARCR) surgery with associated pathology (CPT code 29827 + associated codes)
3. Be scheduled for ARCR surgery for primary repair
4. Be scheduled for ARCR surgery to be performed at Roanoke Ambulatory Surgery Center (RASC) by a surgeon participating in the study
5. Is willing to fill out the pain diary
6. Is able to read, understand, and sign the informed consent document
7. Is able to read and understand the patient-reported measures that will be collected via the pain diary and phone calls

Exclusion Criteria:

1. American Society of Anesthesiologists (ASA) status IIIb or greater.

   ASA status III is characterized by:
   * A patient with severe systemic disease, e.g., Substantive functional limitations; One or more moderate to severe diseases. Examples include (but not limited to): poorly controlled DM or HTN, COPD, morbid obesity (BMI ≥40), active hepatitis, alcohol dependence or abuse, implanted pacemaker, moderate reduction of ejection fraction, ESRD undergoing regularly scheduled dialysis, premature infant PCA < 60 weeks, history (>3 months) of MI, CVA, TIA, or CAD/stents.

   According to Dr. TK Miller and Anesthesiologists at RASC, there is an unwritten standard that patients characterized as ASA status III that have stable, long term disease can be operated on at free-standing ambulatory surgery centers. Broken down into ASA IIIa and ASA IIIb.
   * ASA IIIa represents ASA status III patients that are assessed by anesthesia and deemed stable enough to operate on at a free-standing ambulatory surgery center.
   * ASA IIIb represents ASA status III patients that are assessed by anesthesia and deemed not stable enough to operate on at a free-standing ambulatory surgery center.

   Examples of individuals that would classify as ASA IIIa include:
   * Someone who has a history of longstanding diabetes that is well managed.
   * Someone who is status post cardiac stent(s) and has had no chest pain or angina since the stents have been placed and has been cleared by their cardiologist to go back to full activity.

   Examples of individuals that would classify as ASA IIIb include:
   * Someone who has a history of longstanding diabetes that is poorly managed.
   * Someone who is status post cardiac stent(s) and has had chest pain or angina since the stents have been placed and has not been cleared by their cardiologist to go back to full activity.
2. Currently pregnant
3. Documented opioid use within 30 days prior to surgery
4. Revision ARCR surgery
5. Currently taking opioid medication for chronic pain management
6. History of documented substance abuse or related disorders
7. Currently enrolled or planning to enroll in another clinical trial during this study that would affect the outcome of this study
8. Allergic reactions to amide anesthetics
9. Neurologic deficit or disability involving the surgical extremity
10. Unwilling or unable to consent
11. History of cognitive or mental health status that would interfere with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Total Opioid Use | 6 week
  Total opioid pills consumed, converted to milligram of morphine equivalents (MME)
Duration of Opioid Use | Total 6 week duration of study
  How long the patients took opioid medications for postoperatively (in hours)
NRS Pain Scores | Total 6 week duration of study
  Pain scores on the Numerical Rating Scale, 1-10 with 1 being no pain and 10 being the worst pain imaginable
IBPS Pain Scores | Total 6 week duration of study
  Pain scores on our Intervention Based Pain Scale, proprietary scale developed by Dr. TK Miller at Carilion Clinic. Patient has 6 options to choose from (unnumbered), that will be assigned a numeric value upon analysis. Scale ranges from 1-6, with lower scores representing more manageable (less severe) pain and higher scores representing less manageable (more severe) pain.

SECONDARY OUTCOMES:
Duration of Nerve Block | Within 5 days postoperatively
  How long until patients regained sensation in the affected limb (in hours)
Patient Satisfaction via Likert scale | 2 weeks postoperatively
  Patient satisfaction regarding their pain control on a Likert scale from 1-5 (very unsatisfied, unsatisfied, neither satisfied or unsatisfied, satisfied and very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas K Miller, MD, Principal Investigator — Section Chief, Sports Medicine, Carilion Clinic
Locations (1):
- Carilion Clinic Institute for Orthopaedics and Neurosciences, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No